CLINICAL TRIAL: NCT05557266
Title: Differential Effectiveness of Two Recovery Strategies at Work, Based on Mindfulness and Physical Exercise, on Levels of Job Stress, Inmunoglobuline A, and Cortisol. A Randomized Controlled Trial
Brief Title: Two Recovery Strategies at Work, Based on Mindfulness and Physical Exercise, on Levels of Stress and Biological Measures
Acronym: ERME2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment. The number of interested people did not allow reaching the necessary sample size.
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Miguel Ángel Santed Germán, PhD, Clinical Psychologist and Professor, Universidad Nacional de Educación a Distancia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PID2019-110490RB-I00 (2)
Record Dates: First submitted 2022-09-21; First posted 2022-09-27 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Mental Health Wellness
Keywords: mindfulness; physical exercise; meditation; mental health; stress; recovery; inmunoglobulin A; cortisol
MeSH Terms: conditions — Motor Activity; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of three groups is proposed, with pretest, posttest and three follow-ups at 1,3, and 6 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of trial participants and care providers is not possible because of obvious differences between the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based intervention (MBI) (Experimental): A 8-week mindfulness-based intervention. From 15 to 30 minutes of practice per session, three times/week through audio guided meditations.
  Interventions: Behavioral: Mindfulness-based intervention
- Physical exercise (PE) (Active Comparator): A 8-week physical exercise intervention. From 15 to 30 minutes of practice per session, three times/week through workout videos.
  Interventions: Behavioral: Physical exercise
- Wait list (WL) (No Intervention): The participants will continue their work activity as usual. This arm will be invited to a mindfulness training once the study finished.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — An mindfulness instructor will conduct meditations lasting 15 to 30 minutes. The first day of each week the intervention will be given in streaming and the rest of the days the participants will have audio files designed ad hoc with the practice of the week so they can do it individually at home.
  Arms: Mindfulness-based intervention (MBI)
Behavioral: Physical exercise — An aerobic and fitness trainer will conduct aerobic exercise lasting 15 to 30 minutes. The first day of each week the intervention will be given in streaming and the rest of the days the participants will have video files designed ad hoc with the practice of the week so they can do it individually at home.The intensity of the chosen exercise will be moderate, maintaining between 120-140 beats per minute.
  Arms: Physical exercise (PE)

SUMMARY:
The present study aims to compare the differential effects of mindfulness meditation (MBI) and physical exercise (PE) on different stress and health variables (self-report means and IgA and cortisol levels). A randomized controlled trial of three groups is proposed, with pretest, posttest and three follow-ups at 1, 3 and 6 months that would be developed among the Guardia Civil (Spanish military police) office staff.

DETAILED DESCRIPTION:
Recovery from fatigue and daily work stress involves mentally disconnecting from work. To achieve this disconnection (or psychological detachment), research has shown that engaging in a variety of interesting and motivating activities for individuals after the workday allows them to achieve this disconnected state of mind and, consequently, facilitates recovery from work. Previous research has shown that two of the most effective recovery activities are physical exercise (PE) and mindfulness meditation (MBI), although the results on the differential effects of the two are not conclusive (Karabinski et al, 2021; Steed et al., 2021; Wendsche et al., 2021).

Thus, the present study aims to compare the differential effects of MBI and PE on different stress and health variables (self-report means and IgA and cortisol levels). A randomized controlled trial of three groups is proposed, with pretest, midtest, posttest and three follow-ups at 1, 3 and 6 months that would be developed among the Guardia Civil (Spanish military police) office staff (N ≥ 150). An MBI, an aerobic PE program and an inactive control / waiting list (LE) condition will be contrasted.

The dependent variables considered are: 1) recovery experiences; 2) perceived stress; 3) general health; 4) job satisfaction; 5) work performance; 6) positive and negative affect; 7) daily states of fatigue, stress, psychological distancing, mindfulness, and sleep; 8) IgA levels in saliva; 9) cortisol levels in saliva.

The intervention program is structured for two months, during which the two intervention groups will carry out their recovery strategy (MBI or PE), starting and increasing the practice 5 minutes every two weeks. The control group will continue as usual.

The investigators believe that this study is a quasi-pioneering initiative because of its theme, uses a robust methodology, and will have an important scientific-technical impact. The importance of the topic addressed in terms of health and business productivity is associated with important contributions in terms of knowledge transfer to companies and society in general.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* To be a full-time worker (≥35 hours/week).

Exclusion Criteria:

* Currently practicing any type of meditation regularly.
* Currently practicing physical activity (aerobic or anaerobic) more than once a week.
* To have a physical or mental illness that prevents moderate exercise or mindfulness practice.
* Very low self-perceived work load, responsability, stress levels.
* To take medication that interferes with salivary inmunoglobulin A (SIgA), i.e., pharmacological treatment that can influence the psychological state.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Salivary Immunoglobulin A (SIgA) | Baseline 1 week before treatment, Pre-treatment the week the interventions begin, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up
  Biological measures. Salivary IgA levels as a biomarker of mucosal inmunity. Salivary IgA levels as a biomarker of mucosal inmunity
Change in Salivary cortisol with five points data | Baseline 1 week before treatment, Pre-treatment the week the interventions begin, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up
  Biological measures. Salivary cortisol levels as a biomarker of stress
Change in General Health with six time points data. | Baseline 1 week before treatment, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up, 3-months follow-up, and 6-months follow-up
  The General Health Questionnaire (GHQ-12) consists of 12 items. It is a unidimensional measure of psychological distress. It is answered on a Likert-type scale from 1 to 4 (1 = Never and 4 = Always). The score was used to generate a total score ranging from 0 to 36.
Change in stress with six time points data. | Baseline 1 week before treatment, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up, 3-months follow-up, and 6-months follow-up
  A single item was used: Stress refers to a person's situation when they feel tense, restless, nervous, or anxious, or are unable to sleep at night because their mind is constantly preoccupied with work-related issues. Please indicate the extent to which you currently feel this type of stress. It has five possible responses on a Likert-type scale from 1 to 5 (being 1 nothing and 5 a lot)
Change in Affective Job Satisfaction with six time points data. | Baseline 1 week before treatment, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up, 3-months follow-up, and 6-months follow-up
  The Brief Index of Affective Job Satisfaction (BIAJS)-Spanish version (BIAJS) consists of 7 items. It is an overall measure of affective job satisfaction. It measures satisfaction in five facets: promotion, co-workers, work itself, supervision and salary. It is answered on a Likert-type scale from 1 to 5 (1 = Strongly disagree and 5 = Strongly agree).
  The score was used to generate a total score ranging from 7 to 35.
Change in Need for Recovery with six time points data. | Baseline 1 week before treatment, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up, 3-months follow-up, and 6-months follow-up
  The Need for Recovery (NFR) Scale consists of 9 items. It facilitates the understanding of the factors that can lead to sustainable working and employability. It is answered on a Likert-type scale from 1 to 5 (1 = Never and 5 = Always).
  The score was used to generate a total score ranging from 1 to 100.Our research team will carry the validation of the Spanish version of NFR.
Change in Individual Work Performance with six time points data. | Baseline 1 week before treatment, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up, 3-months follow-up, and 6-months follow-up
  The Individual Work Performance Questionnaire (IWPQ)-Brief Spanish version (IWPQ) has 18 items. It measures the three main dimensions of job performance: task performance, contextual performance, and counterproductive work behavior. It is answered on a Likert-type scale from 1 to 5 (1 = Never or Seldom and 5 = Always or Often). The score was used to generate a total score ranging from 18 to 90.
Change in Positive and Negative Affect with six time points data. | Baseline 1 week before treatment, Mid-treatment 5 weeks from baseline, Post-treatment 9 weeks from baseline, 1-month follow-up, 3-months follow-up, and 6-months follow-up
  The PANAS Scales of Positive and Negative Affect (PANAS) - Spanish version has 20 items. It is the most widely used scale of affectivity. It has two dominant dimensions, positive affect (10 items) and negative affect (10 items) It is answered on a Likert-type scale from 1 to 5 (1 = Very slightly or Not at all and 5 = Extremely). The score was used to generate a total score ranging from 20 to 100.

SECONDARY OUTCOMES:
Change in Fatigue (single-item measure from the Single-Item Fatigue Measure) | 4 days per week during the 8-week interventions
  Single-Item on fatigue level:" Indicate what level of fatigue you felt today". The response is rcorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Psychological distancing (item n. 3 from the Recovery Experience Questionnaire). | 4 days per week during the 8-week interventions
  Single-Item on Psychological distancing level: "After work, I have been able to "disconnect". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Sleep (item n. 6 from the Pittsburg Sleep Quality Index). | 4 days per week during the 8-week interventions
  Single-Item on Sleep: "How did you sleep last night?". The responses are articulated on a Likert-type scale from 1 to 5
  (1 = very bad and 5 = very good)
Change in Work stress (single-item measure from the Single-item Measure of Stress Symptoms). | 4 days per week during the 8-week interventions
  Single-Item on work stress: "Indicate the extent to which you have felt stressed, tense, nervous, or anxious today". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Mindfulness (item n. 3 from the Five Facets Mindfulness Questionnaire). | 4 days per week during the 8-week interventions
  Single-Item on attention: "Today it has been difficult for me to be attentive to what required my attention at all times".
  The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Santed, PhD, Principal Investigator — UNED
Locations (1):
- Raquel Ruiz Iñiguez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided